CLINICAL TRIAL: NCT01431976
Title: A Multi-center, Uncontrolled, Open-label, Evaluation of Lamotrigine Monotherapy on Newly Diagnosed Typical Absence Seizures in Children and Adolescents
Brief Title: Clinical Study of Lamotrigine to Treat Newly Diagnosed Typical Absence Seizure in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115377
Record Dates: First submitted 2011-09-01; First posted 2011-09-12 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lamotrigine (Experimental): No comparison
  Interventions: Drug: Lamictal

INTERVENTIONS:
Drug: Lamictal — No comparison

SUMMARY:
This is a multi-center, uncontrolled, open-label study to evaluate the efficacy and safety of lamotrigine monotherapy on newly diagnosed typical absence seizure in children and adolescents in Japan and South Korea.

The study period is composed the baseline, fixed escalation phase, escalation phase, maintenance phase, taper phase, and post study examination. During the fixed escalation phase, the investigational product is administered at 0.3 mg/kg/day for 2 weeks (Week 1 to 2), followed by 0.6 mg/kg/day for 2 weeks (Week 3 to 4). Subjects thereafter visit the clinic once every 1 to 2 weeks during the escalation phase to increase the dose by 0.6 mg/kg/day up to a maximum of 10.2 mg/kg/day or 400 mg/day (whichever was less) until patients are confirmed to be seizure-free by HV tests for clinical signs. After seizure free is confirmed by HV-clinical signs, the dose is increased by one level and HV-EEG (electroencephalography) test (first test) is assessed at the next visit. If seizure free is observed by HV-EEG, the same dose is administered. Thereafter, HV-EEG (second test) is assessed at the next visit and if seizure free is confirmed again, the subjects enter the 12-week maintenance phase. During the maintenance phase, patients visit the clinic once every 4 weeks. The dose can be adjusted as necessary within the range of 1.2 to 10.2 mg/kg/day or 400 mg/day (whichever was less) taking into account the status of seizures and the safety. The investigational product is administered once daily (in the evening). However, if the number of tablets is large, twice-daily administration (in the morning and evening) is also allowed. After the completion of maintenance phase, subjects who have responded to lamotrigine without tolerability issues are eligible to enter the extension phase of the study if clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Target disease: Subjects with newly diagnosed and untreated typical absence seizure which is classifiable by the International Classification of Seizures.
2. Diagnosis of typical absence seizures is established by at least one of two 4-minute hyperventilation tests as supported by clinical signs and EEG findings.

   The following criteria will be used to define a typical absence seizure on the EEG: a discharge of generalized spike-and-wave or multiple spike-and-wave activity lasting ≥3 seconds during the awake state. The frequency of the spike-and-wave should be between 2.5-4.5 Hz.
3. Age (at the time of obtaining consent):

   * 2 to 15 years of age in Japan
   * 2 to 12 years of age in South Korea
4. Subjects must weigh at least 7 kg
5. Outpatients
6. Parent/guardian must have given written informed consent. Subjects who are intellectually able to understand the concepts and procedures of the protocol must give assent by also signing the consent.
7. Gender: Male or female
8. QTc<450 millisecond (msec) or <480msec for subjects with Bundle Branch Block - values based on either single ECG values or triplicate ECG averaged QTc values obtained over a brief recording period.

Exclusion Criteria:

1. Subjects with partial seizure or generalized seizures other than typical absence.
2. Subjects with a history of rash associated with other treatment.
3. Subjects with any clinically significant chronic cardiac, renal, or hepatic medical condition. Any patient with these conditions will be excluded from the study even if these conditions are being controlled with chronic therapy.
4. Subjects with an acute or chronic illness likely to impair drug absorption, distribution, metabolism or excretion or with any unstable physical symptoms likely to require hospitalization during participation in the study.
5. Subjects with a psychiatric disorder requiring medication, or who had psychiatric conditions in the past that was both judged to be severe and required hospitalization.
6. Subjects with an acute or progressive neurological disorder or an organic disease.
7. Subjects with currently taking any psychoactive drugs to treat hyperactivity disorder or attention deficit disorder.
8. Subjects with an unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
9. Female subjects who are pregnant or lactating, who may be pregnant, or who plan for pregnancy during the study.
10. Children in foster care: A child who has been placed under the control or protection of an agency, organisation, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. This can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The definition of a child in care does not include a child who is adopted or who has an appointed legal guardian.
11. Subjects taking inducers of lamotrigine glucuronidation (i.e., rifampicin, lopinavir/ritonavir), atazanavir/ritonavir, risperidone, oral contraceptives or hormone drug which includes estrogen.
12. Subjects having participated in other clinical study in the past 3 months before the start of investigational product.
13. Subjects who have active suicidal plan/intent or have had active suicidal thoughts in the past 3 months before the start of investigational product or who have history of suicide attempt in the last 1 year before the start of investigational product or more than 1 lifetime suicide attempt.
14. Subjects whom the investigator (or subinvestigator) considers ineligible for the study.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- Japan (10):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Yasumoto S, Shimizu M, Sato K, Kurata A, Numachi Y. Lamotrigine monotherapy for newly diagnosed typical absence seizures in children: A multi-center, uncontrolled, open-label study. Brain Dev. 2016 Apr;38(4):407-13. doi: 10.1016/j.braindev.2015.10.007. Epub 2015 Oct 27. PMID 26518979
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 115377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115377 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with newly diagnosed and untreated typical absence seizure; aged 2-15 years in Japan, 2-12 years in South Korea at the time of obtaining consent; weighing at least 7 kilograms (kg); without partial seizure or generalized seizures other than typical absence; and without a history of rash associated with other treatment were enrolled.
Pre-assignment Details: The study consisted of an Escalation Phase (EP), a 12-week (W) Maintenance Phase (MP), a >=2-week Taper Phase, and post-study examination within 1-4 weeks after the last dose of lamotrigine. Participants could have entered the Extension Phase (ExP) until approval for this indication or until 24 months after the Last Subject Last Visit in the MP.
Groups:
- Lamotrigine: In the EP, lamotrigine 0.3 milligrams per kilogram per day (mg/kg/day) was administered orally once daily from Week W1 to W2, and 0.6 mg/kg/day from W3 to W4. From W5, the dose was escalated by 0.6 mg/kg/day once every 1 or 2 weeks, up to a maximum of 10.2 mg/kg/day or 400 mg/day, whichever was less (WWL), until a seizure-free (SF) status was confirmed by hyperventilation (HV)-clinical signs. After a SF confirmation, the dose was increased by one level and HV-electroencephalography was assessed twice at the same dose level to confirm the SF status. In the MP, the same dose was continued for 12 weeks. An increase/decrease in dose (0.6 mg/kg/day at >=1-week intervals) was allowed within the range of 1.2 to 10.2 mg/kg/day or 400 mg/day, WWL. In the ExP, doses of 1.2 to 10.2 mg/kg/day or 400 mg/day (WWL) were administered based on seizure status/safety. If a dose <1.2 mg/kg/day or >10.2 mg/kg/day or 400 mg/day (WWL) was necessary, the participant was withdrawn from the study.
Period: Overall Study
Arm/Group | Lamotrigine
Started | 20
Completed | 6
Not Completed | 14
Not completed — Adverse Event | 6
Not completed — Lack of Efficacy | 2
Not completed — Met Protocol-defined Stopping Criteria | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Lamotrigine: In the EP, lamotrigine 0.3 mg/kg/day was administered orally once daily from W1 to W2, and 0.6 mg/kg/day from W3 to W4. From W5, the dose was escalated by 0.6 mg/kg/day once every 1 or 2 weeks, up to a maximum of 10.2 mg/kg/day or 400 mg/day, WWL, until a SF status was confirmed by HV-clinical signs. After a SF confirmation, the dose was increased by one level and HV-electroencephalography was assessed twice at the same dose level to confirm the SF status. In the MP, the same dose was continued for 12 weeks. An increase/decrease in dose (0.6 mg/kg/day at >=1-week intervals) was allowed within the range of 1.2 to 10.2 mg/kg/day or 400 mg/day, WWL. In the ExP, doses of 1.2 to 10.2 mg/kg/day or 400 mg/day (WWL) were administered based on seizure status/safety. If a dose <1.2 mg/kg/day or >10.2 mg/kg/day or 400 mg/day (WWL) was necessary, the participant was withdrawn from the study.
Arm/Group | Lamotrigine
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.7 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race/Ethnicity, Customized [Number; unit: participants]
  East Asian Heritage | 3
  Japanese Heritage | 16
  South East Asian Heritage | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Seizure Free as Confirmed by Hyperventilation (HV)-Electroencephalography (EEG) at the End of the Maintenance Phase (MP)
Description: EEG is a diagnostic test for epilepsy. The EEG machine records the brain's electrical activity as a series of waveforms. HV is an activation technique used to provoke seizures during an EEG recording. An approximately 30-minute EEG with HV was performed on participants in a supine position. In the HV test, participants breathed through their mouths deeply and rapidly (at a rate of approximately 20-25 breaths/minute) for 4 continuous minutes using a pin-wheel provided to them.
Time Frame: Week 12 of the Maintenance Phase (up to Study Week 50)
Population: Full Analysis Set (FAS): all participants who took at least one dose of investigational product and contributed data to at least one efficacy measure after the first dosing of investigational product
Measure: Number; unit: Participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 20
Participants | 7
Statistical Analysis 1: Comparison: Lamotrigine; Test type: Superiority or Other; percentage of participants = 35.0, 95% CI 2-sided [15.39 to 59.22]

2. Secondary Outcome: Number of Participants Who Were Seizure Free as Confirmed by HV-EEG at Two Consecutive Visits in the Escalation Phase (EP)
Description: EEG is a diagnostic test for epilepsy. The EEG machine records the brain's electrical activity as a series of waveforms. HV is an activation technique used to provoke seizures during an EEG recording. An approximately 30-minute EEG with HV was performed on participants in a supine position. In the HV test, participants breathed through their mouths deeply and rapidly (at a rate of approximately 20-25 breaths/minute ) for 4 continuous minutes using a pin-wheel provided to them.
Time Frame: Up to Study Week 49
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 20
Participants | 8

3. Secondary Outcome: Number of Participants Who Were Seizure Free as Confirmed by HV-clinical Signs at Each Dose During the Escalation Phase
Description: HV is an activation technique used to provoke seizures. Participants were instructed to breathe through their mouths deeply and rapidly (at a rate of approximately 20-25 breaths/minute) for 4 continuous minutes while sitting using a pin-wheel and were observed for clinical signs of seizures like impairment of consciousness; staring; eye enrollment; eye blinking; chewing movements; hand movement; other automatisms; atonic, tonic, clonic components; autonomic components; or any other signs. During the Escalation Phase, HV-clinical signs were assessed to confirm a status of seizure free. Only participants data available at the analysis time point were analyzed (represented as n=X, X, X in category title).
Time Frame: Up to Study Week 49
Population: FAS. Only those participants given the indicated dose of investigational product were analyzed.
Measure: Number; unit: Participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 20
Participants
  0.6 mg/kg, n=17 | 1
  1.2 mg/kg, n=17 | 1
  1.8 mg/kg, n=16 | 2
  2.4 mg/kg, n=16 | 2
  3.0 mg/kg, n=16 | 2
  3.6 mg/kg, n=15 | 1
  4.2 mg/kg, n=15 | 0
  4.8 mg/kg, n=14 | 4
  5.4 mg/kg, n=14 | 1
  6.0 mg/kg, n=11 | 1
  6.6 mg/kg, n=11 | 0
  7.2 mg/kg, n=9 | 3
  7.8 mg/kg, n=9 | 0
  8.4 mg/kg, n=6 | 2
  9.0 mg/kg, n=6 | 1
  9.6 mg/kg, n=1 | 1

4. Secondary Outcome: Number of Participants Who Were Seizure Free as Confirmed by HV-clinical Signs During Week 4 and Week 8 of the Maintenance Phase
Description: HV is an activation technique used to provoke seizures. Participants were instructed to breathe through their mouths deeply and rapidly (at a rate of approximately 20-25 breaths/minute) for 4 continuous minutes while sitting using a pin-wheel and were observed for clinical signs of seizures like impairment of consciousness; staring; eye enrollment; eye blinking; chewing movements; hand movement; other automatisms; atonic, tonic, clonic components; autonomic components; or any other signs. During the Maintenace Phase, HV-clinical signs were assessed at Visit 1 (Week 4) and Visit 2 (Week 4).
Time Frame: Week 4 and Week 8 of the Maintenance Phase (up to Study Weeks 42 and 46, respectively)
Population: FAS. Only those participants who were dosed with investigational product at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 7
Participants
  Week 4 | 7
  Week 8 | 7

5. Secondary Outcome: Number of Participants Who Were Seizure Free as Confirmed by HV-EEG at Each Assessment Point in the Extension Phase (ExP)
Description: EEG is a diagnostic test for epilepsy. The EEG machine records the brain's electrical activity as a series of waveforms. HV is an activation technique used to provoke seizures during an EEG recording. An approximately 30-minute EEG with HV was performed on participants in a supine position. In the HV test, participants breathed through their mouths deeply and rapidly (at a rate of approximately 20-25 breaths/minute ) for 4 continuous minutes using a pin-wheel provided to them. Only participants data available at the analysis time point were analyzed (represented as n=X, X, X in category title).
Time Frame: Extension Week 12 (Extension Visit 1 [Ext-V1]), every 24 weeks after Ext-V1 and until withdrawal
Population: FAS. Only those participants given the indicated dose of investigational product were analyzed.
Measure: Number; unit: Participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 20
Participants
  Extension Week 12, n=7 | 6 (1.568)
  Extension Week 36, n=7 | 5 (2.114)
  Extension Week 60, n=7 | 6 (0.161)
  Extension Week 84, n=6 | 6 (2.197)
  Extension Week 108, n=6 | 6
  Extension Week 132, n=6 | 6
  Extension Week 156, n=2 | 2

6. Secondary Outcome: Number of Participants Who Were Seizure Free as Confirmed by HV-clinical Signs at Each Assessment Point in the Extension Phase (ExP)
Description: HV is an activation technique used to provoke seizures. Participants were instructed to breathe through their mouths deeply and rapidly (at a rate of approximately 20-25 breaths/minute) for 4 continuous minutes while sitting using a pin-wheel and were observed for clinical signs of seizures like impairment of consciousness; staring; eye enrollment; eye blinking; chewing movements; hand movement; other automatisms; atonic, tonic, clonic components; autonomic components; or any other signs. During the ExP, HV-clinical signs were assessed to confirm a status of seizure free. Only participants data available at the analysis time point were analyzed (represented as n=X, X, X in category title).
Time Frame: Extension Week 24 (Extension Visit 2 [Ext-V2], every 24 weeks after the Ext-V2 and until withdrawal
Population: FAS. Only those participants given the indicated dose of investigational product were analyzed.
Measure: Number; unit: Participants
Arm/Group | Lamotrigine
Number analyzed (Participants) | 20
Participants
  Extension Week 24, n=7 | 5
  Extension Week 48, n=7 | 6
  Extension Week 72, n=7 | 5
  Extension Week 96, n=6 | 6
  Extension Week 120, n=6 | 5
  Extension Week 144, n=4 | 2
  Extension Week 168, n=1 | 1

7. Secondary Outcome: Number of Days With Seizure Episodes Per Week in the Main Study Phase (Fixed Escalation Phase [FEP], Escalation Phase [EP], Maintenance Phase [MP]), and FEP+EP+MP)
Description: Participants were asked to record the seizure codes, seizure duration, and their physical condition in a diary provided. Only participants data available at the analysis time point were analyzed (represented as n=X, X, X in category title)
Time Frame: Up to Study Week 50
Population: FAS
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lamotrigine
Number analyzed (Participants) | 20
Days
  Fixed Escalation Phase, n=20 | 4.93 (1.488)
  Escalation Phase, n=17 | 2.60 (2.060)
  Maintenance Phase, n=8 | 0.06 (0.161)
  FEP+EP+MP, n=20 | 2.98 (1.976)

8. Secondary Outcome: Number of Days With Seizure Episodes Per Week in the Extension Phase (ExP) Overall
Description: Participants were asked to record the seizure codes, seizure duration, and their physical condition in a diary provided.
Time Frame: Extension Week 12 (Extension Visit 1 [Ext-V1], every 12 week after Ext-V1 and until withdrawal
Population: FAS. Only those participants given the indicated dose of investigational product were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Lamotrigine
Number analyzed (Participants) | 7
Days | 0.03 (0.048)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from study medication start until the end of treatment (up to Study Week 50) (EP, MP, and ExP).
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who had taken at least one dose of investigational product.
Arm/Group | Lamotrigine
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 17/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lamotrigine (N=20)
Bronchitis (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 5
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Pneumonia mycoplasmal (Infections and infestations) | 1
Scarlet fever (Infections and infestations) | 1
Varicella (Infections and infestations) | 2
Adenovirus infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Otitis media acute (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 2
Rash (Skin and subcutaneous tissue disorders) | 6
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 3
Chillblains (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 4
Psychomotor hyperactivity (Nervous system disorders) | 1
Febrile convulsion (Nervous system disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Proteinuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pain (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.